CLINICAL TRIAL: NCT03216460
Title: Evaluating Glucose Control in Patients With Type 1 Diabetes Under Free-living Conditions With the Insulet Automated Glucose Control System: IDE3
Brief Title: Insulet Artificial Pancreas Free-Living IDE3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insulet Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IDE3
Record Dates: First submitted 2017-07-01; First posted 2017-07-13 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Type1 Diabetes Mellitus
Keywords: T1D, Omnipod
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This study is a single-arm, multi-center, observational clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Supervised Free-Living (Other): Subjects will undergo a 7±1 day outpatient, standard therapy phase during which sensor and insulin data will be collected. Subjects or their caregivers will manage their diabetes at home per their usual routine using the study CGM and remain on current MDI or pump therapy. This will be followed by a 5-day/4-night or from approximately 48 to 72 hours for children ages 2.0-5.9 years, hybrid closed-loop phase conducted in a supervised hotel/rental house setting, where subjects will participate in specific setpoint challenges, meal challenges, and exercise
  Interventions: Device: Insulet automated glucose control system

INTERVENTIONS:
Device: Insulet automated glucose control system — Insulet AP (artificial pancreas) system, using the Omnipod® insulin management system, Dexcom G4Share® AP System and personalized model predictive control algorithm.

SUMMARY:
Subjects will undergo a 7±1 day outpatient, standard therapy phase during which sensor and insulin data will be collected. Subjects or their caregivers will manage their diabetes at home per their usual routine using the study CGM and remain on current MDI or pump therapy. This will be followed by a 5-day/4-night or from approximately 48 to 72 hours for children ages 2.0-5.9 years, hybrid closed-loop phase conducted in a supervised hotel/rental house setting.

DETAILED DESCRIPTION:
The study schedule will consist of a standard therapy data collection week followed by a hybrid closed-loop phase.

Subjects will undergo a 7±1 day outpatient, standard therapy phase during which sensor and insulin data will be collected. Subjects or their caregivers will manage their diabetes at home per their usual routine using the study CGM and remain on current MDI or pump therapy. This will be followed by a 5-day/4-night or from approximately 48 to 72 hours for children ages 2.0-5.9 years, hybrid closed-loop phase conducted in a supervised hotel/rental house setting.

The hybrid closed-loop phase will begin prior to lunch on Study Day 1.

During the hybrid closed-loop phase, subjects will participate in specific setpoint challenges, meal challenges, and exercise.

Hybrid closed-loop will be discontinued approximately 5 hours after breakfast time on Study Day 5. Subjects will be asked to complete a post-study questionnaire regarding their experience with the system. Subjects will be discharged home when stable and all discharge criteria are met. Subjects will consume a snack or meal after discontinuation of hybrid closed-loop before they leave the study site.

ELIGIBILITY:
Inclusion Criteria:

1. Age at time of consent 2.0-85 years
2. Individuals aged ≥6.0 must be diagnosed with type 1 diabetes for at least one year. Preschool children aged 2.0-5.9 years must be diagnosed with type 1 diabetes for at least 6 months. Diagnosis is based on investigator's clinical judgment.
3. A1C <10% at screening
4. Currently using U-100 rapid-acting insulin analogs with insulin pump or receiving multiple daily injections suitable for conversion to pump therapy for at least 3 months prior to study start
5. Willing to use the study CGM device for the duration of the study
6. Willing to use the Omnipod® Insulin Management System during the study
7. Willing to perform all fingerstick BG testing with the study-approved glucose meter at the frequency specified in the study protocol or per investigator discretion
8. Willing to participate in setpoint and meal challenges
9. Willing to use carbohydrate counting for determination of meal boluses
10. Willing to participate in moderate intensity exercise for at least 30 minutes per day
11. Willing to refrain from use of acetaminophen and supplemental vitamin C (>2000 mg/daily) for the entire duration of participation in the study
12. Willing and able to sign the Informed Consent Form (ICF) and/or has a parent/guardian willing and able to sign the ICF. Assent will be obtained from pediatric and adolescent subjects per State requirements.

Exclusion Criteria:

1. One or more episodes of severe hypoglycemia requiring emergency room (ER) visit or hospitalization within the past 6 months
2. One or more episodes of diabetic ketoacidosis requiring ER visit or hospitalization within the past 6 months
3. Planning to start a non-insulin anti-diabetic medication during the study. If on non-insulin medication, dose must be stable in the previous 30 days.
4. Using a basal insulin with a usual duration of insulin action > 36 hours
5. Pregnant or lactating, or is a woman of childbearing potential and not on acceptable form of birth control (acceptable includes abstinence, condoms, oral/injectable contraceptives, IUD or implant)
6. Dermatological conditions at the proposed sensor/pump wear sites that in the investigator's opinion could preclude ability to wear the Pod and/or the Dexcom sensor
7. Current or known history of coronary artery disease that is not stable with medical management, including unstable angina, or angina that prevents moderate exercise despite medical management, or a history of myocardial infarction, percutaneous coronary intervention, or coronary artery bypass grafting within the previous 12 months. Abnormal electrocardiogram consistent with increased risk of arrhythmia, ischemia, or prolonged QT interval (> 440 ms). Electrocardiogram is only required for subjects >50 years old or with diabetes duration >20 years.
8. Stroke
9. Known history of seizure disorder
10. Known history of adrenal insufficiency
11. Current renal or hepatic disease
12. Untreated or unstable hypothyroidism or celiac disease (per investigator's judgment)
13. Currently undergoing cancer treatment
14. Currently undergoing systemic treatment with steroids or immunosuppressive medication
15. Known history of any chronic infections that would interfere with participation in the study or place study personnel at undue risk due to blood-borne contaminants
16. Current illness that would interfere with participation in the study
17. Untreated or inadequately treated mental illness
18. Current alcohol abuse per investigator's judgment
19. Electrically-powered implants that may be susceptible to RF interference
20. Currently participating in another clinical study using an investigational drug or device
21. Recent (within the preceding 30 days) participation in a clinical study using an investigational drug
22. Unable to follow the clinical protocol for the duration of the study or is otherwise deemed unacceptable to participate in the study per the investigator's clinical judgment.

Ages: 2 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Percentage of time in hypoglycemic range (defined as < 70 mg/dL) | 96 hours
Percentage of time in hyperglycemic range (defined as ≥ 250 mg/dL) | 96 hours

SECONDARY OUTCOMES:
Mean Glucose | 96 hours
Percentage of time < 50 mg/dL | 96 hours
Percentage of time < 54 mg/dL | 96 hours
Percentage of time < 60 mg/dL | 96 hours
Percentage of time > 180 mg/dL | 96 hours
Percentage of time ≥ 300 mg/dL | 96 hours
Percentage of time between 70-180 mg/dL | 96 hours
Percentage of time between 70-140 mg/dL | 96 hours
Standard deviation | 96 hours
  Using CGM measurements, the Standard deviations will be reported for the entire hybrid closed-loop phase overall, as well as separately during the day (0700 - 2259h) and during the night (2300 - 0659h).
Coefficient of variation | 96 hours
  Using CGM measurements, the Coefficient of variation will be reported for the entire hybrid closed-loop phase overall, as well as separately during the day (0700 - 2259h) and during the night (2300 - 0659h).

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Stanford University, Palo Alto, California
  - University of Colorado Denver, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No